CLINICAL TRIAL: NCT06085950
Title: Transcranial Ultrasonic Stimulation in Treatment-resistant Depression: an Open-label Pilot Trial
Brief Title: Transcranial Ultrasonic Stimulation in Treatment-resistant Depression : an Open-label Pilot Trial
Acronym: StimulUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D21-P020
Record Dates: First submitted 2023-09-12; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcranial Ultrasonic Stimulation with Personalized Acoustic Lens (Experimental): Low-intensity transcranial focused ultrasound stimulation of deep brain target, using a personalized acoustic lens to correct the aberrations induced by the skull
  Interventions: Device: Transcranial Ultrasonic Stimulation prototype

INTERVENTIONS:
Device: Transcranial Ultrasonic Stimulation prototype — Transcranial Ultrasonic Stimulation prototype delivers personalized low-intensity ultrasound stimulation

SUMMARY:
The primary objective of this study is to optimize the protocol for the TUS administration in patients with TRD while gaining an initial impression of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years,
* Diagnosis of major depressive episode (MDE) as part of major depressive disorder as defined by DSM-5 criteria
* Severe MDE (HDRS-17> 20)
* Drug resistance to at least two well-conducted antidepressant treatment lines
* With stable antidepressant treatment for at least 4 weeks before inclusion
* Benefiting from a social security scheme
* Having given their consent to participate

Exclusion Criteria:

* Psychiatric history other than a mood disorder
* Neurological history, including epilepsy and intracerebral calcifications
* History of substance use disorder other than tobacco
* Contraindication to brain MRI (pacemaker, neurostimulator, injury from metallic shine, …)
* Compulsory psychiatric care
* Protected adults, people under legal safeguard
* Pregnant or breastfeeding woman
* Women of childbearing age who do not have a negative pregnancy test and are not using contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-05-13 (Estimated); Study Completion 2024-06-12 (Estimated)

PRIMARY OUTCOMES:
Percent change in the Montgomery-Åsberg Depression Scale (MADRS) score from baseline to primary endpoint | Pre-treatment and Day 5 from start of intervention
  MADRS is a ten item diagnostic questionnaire used to measure the severity of depressive symptoms in patients with mood disorders. Scale range - 0 to 60 with higher score indicative of greater depressive symptomology.

SECONDARY OUTCOMES:
Incidence of serious adverse reactions according to the Common Terminology Criteria for Adverse Events (CTCAE) scale | Day 1 to Day 35 from start of intervention
  CTCAE are a set of criteria for the standardized classification of adverse effects
Percent change in the Montgomery-Åsberg Depression Scale (MADRS) | Pre-treatment and Day 1, Day 2, Day 3, Day 4, Day 5, Day 12 ± 2, Day 19 ± 2, Day 26 ± 2, Day 33 ± 2 from start of intervention
  MADRS is a ten item diagnostic questionnaire used to measure the severity of depressive symptoms in patients with mood disorders. Scale range - 0 to 60 with higher score indicative of greater depressive symptomology.
Percent change in the Hamilton Rating Scale for Depression (HDRS-17) | Pre-treatment and Day 1, Day 2, Day 3, Day 4, Day 5, Day 12 ± 2, Day 19 ± 2, Day 26 ± 2, Day 33 ± 2 from start of intervention
  HDRS-17 is a 17 item questionnaire used to score the severity of depression. Scale range - 0 to 52 with higher score indicative of greater depressive symptomology.
Percent change in the Hamilton Rating Scale for Depression (HDRS-6) | Pre-treatment and Day 1, Day 2, Day 3, Day 4, Day 5, Day 12 ± 2, Day 19 ± 2, Day 26 ± 2, Day 33 ± 2 from start of intervention
  HDRS-6 is a 6 item questionnaire used to score the severity of depression. Scale range - 0 to 22 with higher score indicative of greater depressive symptomology.
Percent change in the Inventory of Depressive Symptomatology (IDC-C) | Pre-treatment and Day 1, Day 2, Day 3, Day 4, Day 5, Day 12 ± 2, Day 19 ± 2, Day 26 ± 2, Day 33 ± 2 from start of intervention
  IDS-C is a 30 item questionnaire used to score the severity of depression. Scale range - 0 to 90 with higher score indicative of greater depressive symptomology.
Percent change in the Quick Inventory of Depressive Symptomatology (QIDS-SR) | Pre-treatment and Day 1, Day 2, Day 3, Day 4, Day 5, Day 12 ± 2, Day 19 ± 2, Day 26 ± 2, Day 33 ± 2 from start of intervention
  QIDS-SR is a 16 item self-administered questionnaire used to score the severity of depression. Scale range - 0 to 27 with higher score indicative of greater depressive symptomology.
Assess the changes in functional connectivity of sgACC after TUS | Pre-treatment and Day 7 from start of intervention
  Comparison of functional connectivity of subgenual cingulate cortex through resting state imaging analysis before / after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Sainte-Anne, Paris, France

REFERENCES:
- [Derived] Attali D, Tiennot T, Manuel TJ, Daniel M, Houdouin A, Annic P, Dizeux A, Haroche A, Dadi G, Henensal A, Moyal M, Le Berre A, Paolillo C, Charron S, Debacker C, Lui M, Lekcir S, Mancusi R, Gallarda T, Sharshar T, Sylla K, Oppenheim C, Cachia A, Tanter M, Aubry JF, Plaze M. Deep transcranial ultrasound stimulation using personalized acoustic metamaterials improves treatment-resistant depression in humans. Brain Stimul. 2025 May-Jun;18(3):1004-1014. doi: 10.1016/j.brs.2025.04.018. Epub 2025 Apr 29. PMID 40311843